CLINICAL TRIAL: NCT04372433
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Intravenously Administered IO-202 and IO-202 + Azacitidine ± Venetoclax in Acute Myeloid Leukemia (AML) Patients With Monocytic Differentiation and in Chronic Myelomonocytic Leukemia (CMML) Patients
Brief Title: IO-202 as Monotherapy and IO-202 Plus Azacitidine ± Venetoclax in Patients in AML and CMML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune-Onc Therapeutics (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IO-202-CL-001
Record Dates: First submitted 2020-04-20; First posted 2020-05-04 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: AML With Monocytic Differentiation; CMML
Keywords: Monocytic
MeSH Terms: interventions — Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation of IO-202 (Experimental): Dose cohorts treated with intravenous (IV) IO-202 monotherapy in ascending doses.
  Interventions: Biological: IO-202
- Dose Escalation of IO-202 Plus Azacitidine (Experimental): AZA Dose cohorts treated with intravenous (IV) IO-202 in ascending doses plus Azacitidine (IV or SC) on days 1-7 of each 28-day cycle.
  Interventions: Biological: IO-202 and Azacitidine
- Dose Expansion of IO-202 plus Azacitidine AML (Experimental): To enroll high LILRB4 expression monocytic AML patients refractory to or relapsed after available therapies known to be active in AML.
  Interventions: Biological: IO-202 and Azacitidine
- Dose Expansion of IO-202 plus Azacitidine CMML (Experimental): To enroll hypomethylating-agent naive CMML patients.
  Interventions: Biological: IO-202 and Azacitidine
- Dose Expansion of IO-202 plus Azacitidine + Venetoclax (Ven) (Experimental): To enroll newly diagnosed high LILRB4 expression AML patients who are unfit for intensive induction chemotherapy.
  Interventions: Biological: IO-202 and Azacitidine + Venetoclax

INTERVENTIONS:
Biological: IO-202 — IO-202 as monotherapy
  Arms: Dose Escalation of IO-202
Biological: IO-202 and Azacitidine — IO-202 and azacitidine combination therapy
  Other Names: IO-202 and AZA
  Arms: Dose Escalation of IO-202 Plus Azacitidine; Dose Expansion of IO-202 plus Azacitidine CMML
Biological: IO-202 and Azacitidine + Venetoclax — IO-202 and azacitidine + venetoclax combination therapy
  Other Names: IO-202 and AZA + Ven
  Arms: Dose Expansion of IO-202 plus Azacitidine + Venetoclax (Ven)
Biological: IO-202 and Azacitidine — IO-202 and azacitidine combination therapy
  Other Names: IO-202 and AZA
  Arms: Dose Expansion of IO-202 plus Azacitidine AML

SUMMARY:
To assess safety and tolerability at increasing dose levels of IO-202 in successive cohorts of participants with AML with monocytic differentiation and CMML in order to estimate the maximum tolerated dose (MTD) or maximum administered dose (MAD) and select the recommended Phase 2 dose (RP2D)

DETAILED DESCRIPTION:
This is a Phase 1, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Intravenously Administered IO-202 and IO-202 + Azacitidine ± Venetoclax in Acute Myeloid Leukemia (AML) Patients with Monocytic Differentiation and in Chronic Myelomonocytic Leukemia (CMML) Patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18.
2. For the Part 1 Dose-Escalation Phase, patients must be diagnosed with the following:

   1. Relapsed or refractory AML with myelomonocytic or monoblastic/monocytic differentiation according to the World Health Organization 2016 criteria and has failed treatment with available therapies known to be active for AML.
   2. Relapsed or refractory CMML and has failed treatment with available therapies known to be active for CMML
3. Part 2 Expansion Phase:

   1. Relapsed or refractory LILRB4high AML with myelomonocytic or monoblastic/monocytic differentiation and has failed treatment with available therapies known to be active for AML.
   2. Hypomethylating-agent naive CMML regardless of LILRB4 expression levels.
   3. Newly diagnosed high LILRB4 expression monocytic AML patients considered to be ineligible for standard induction therapy.
4. Patients must be amenable to serial BM aspirates/biopsies and peripheral blood sampling during the study.
5. Patients must be able to understand and willing to sign an informed consent. A legally authorized representative may consent.
6. Patients must have an ECOG performance status of 0 to 2
7. Patients must have adequate hepatic function
8. Patients must have adequate renal function
9. Patients must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer.
10. Patients must be off systemic calcineurin inhibitors for at least 4 weeks prior to study drug treatment.
11. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy.

Exclusion Criteria:

1. Patients who have previously received a monoclonal antibody therapy targeting LILRB4.
2. Patients who have undergone HSCT within 60 days of the first dose of IO-202.
3. Patients who received systemic anti-cancer therapy or radiotherapy <7 days prior to their first day of study drug administration (Hydroxyurea or leukapheresis is allowed up to 24 hours prior to the first dose.
4. Patients who received an investigational agent <7 days prior to their first day of study drug administration.
5. Patients for whom potentially curative anti-cancer therapy is available.
6. Patients who are pregnant or breastfeeding.
7. Patients with uncontrolled, active infection.
8. Patients with known hypersensitivity to any of the components of the IO-202 formulation.
9. Patients with known pulmonary lesions and/or history of pneumonitis or interstitial lung disease.
10. Active known malignancy.
11. Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF) or left ventricular ejection fraction (LVEF) <40%.
12. Ongoing cardiac dysrhythmias Grade 2 or higher per of NCI CTCAE, Version 5.0, Grade ≥2.
13. Known or suspected hypersensitivity to recombinant proteins.
14. Known active bacterial, viral, and/or fungal infection.
15. Patients with any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol.
16. Patients with clinical signs and/or symptoms suggesting active, uncontrolled central nervous system (CNS) leukemia or known active, uncontrolled CNS leukemia.
17. Patients with immediately life-threatening, severe complications of leukemia.
18. Donor Lymphocyte Infusion within 30 days prior to first IO-202 administration.
19. Current active treatment in another interventional therapeutic clinical study.
20. Chronic systemic corticosteroid treatment with a dose of >10 mg prednisone/day or dose equivalent.
21. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
22. Acute Promyelocytic Leukemia patients or patients with known Philadelphia chromosome (Ph+) positive AML or chronic myelogenous leukemia (CML) blast crisis.
23. Hyperleukocytosis (leukocytes ≥25 x 10e9/L) at first dose of IO-202.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Safety of IO-202 and IO-202 plus azacitidine ± venetoclax as measured by incidence of adverse events. | From first dose of IO-202 to 30 days following last study treatment
  Incidence of adverse events
Safety of IO-202 and IO-202 plus azacitidine ± venetoclax as measured by incidence of adverse events. | From first dose of IO-202 to 30 days following last study treatment
  Severity of adverse events
Tolerability of IO-202 and IO-202 plus azacitidine ± venetoclax as measured by incidence and duration of dose interruptions and dose reductions of study treatment. | From first dose of IO-202 to 30 days following last study treatment
  Incidence dose interruptions and dose reductions

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of IO-202 and IO-202 plus azacitidine ± venetoclax and as defined by maximum plasma concentration (Cmax) | Through study completion, an average of 1 year
  Maximum concentration (Cmax) of IO-202
To characterize the PK of IO-202 and IO-202 IO-202 plus azacitidine ± venetoclax as defined by area under the curve (AUC) | Through study completion, an average of 1 year
  measure area under the curve (AUC) of IO-202
To evaluate the incidence of anti-drug antibodies against IO-202 | Through study completion, an average of 1 year
  Measure anti-drug antibodies in plasma.
To measure rates of response to IO-202 and IO-202 plus azacitidine ± venetoclax | Through study completion, an average of 1 year
  Measure response rates in patients with anti-drug antibodies.

OTHER OUTCOMES:
To correlate target expression with response rates | Through study completion, an average of 1 year
  Statistical correlation levels of target expression on leukemic blasts with response rate
To correlate target expression with rates of adverse events | Through study completion, an average of 1 year
  Statistical correlation of target expression on leukemic blasts with adverse event rates
To evaluate immunophenotype of leukemic blasts after study treatment. | Through study completion, an average of 1 year
  Measure immunophenotype of leukemic blasts from bone marrow aspirates after study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xiang, PhD, Study Director — Immune-Onc Therapeutics
Locations (14):
- United States (14):
  - University California, Davis (117), Davis, California
  - City of Hope (106), Duarte, California
  - University of California, Irvine (107), Irvine, California
  - UCLA, Medical Center Division of Hematology/Oncology (119), Los Angeles, California
  - Stanford University (114), Palo Alto, California
  - University of California, San Francisco (118), San Francisco, California
  - University of Colorado, Anschutz Medical Campus (103), Aurora, Colorado
  - Winship Cancer Institute of Emory University (105), Atlanta, Georgia
  - The University of Chicago (113), Chicago, Illinois
  - Weill Cornell Medical College, New York Presbyterian Hospital (110), New York, New York
  - Cleveland Clinic, Taussig Cancer Institute (111), Cleveland, Ohio
  - Oregon Health and Science University, Center for Hematologic Malignancies (116), Portland, Oregon
  - University of Texas Southwestern, Simmons Comprehensive Cancer Center (104), Dallas, Texas
  - MD Anderson Cancer Center (101), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aribi A, Mannis GN, Madanat YF, Jonas BA, Dunavin N, Roboz GJ, Jeyakumar D, Garcia-Manero G, Liu H, Carraway HE, Saultz JN, Blum W, Schiller G, Huang T, Woodard P, Klencke B, Liao XC, Xiang H, Pollyea DA, DiNardo CD. A phase 1 study of IO-202, an anti-LILRB4 antibody, in chronic myelomonocytic leukemia and acute myeloid leukemia. Blood Neoplasia. 2025 Jun 9;2(4):100126. doi: 10.1016/j.bneo.2025.100126. eCollection 2025 Nov. PMID 40919482